CLINICAL TRIAL: NCT06825065
Title: Acute Effects of Post-Activation Performance Enhancement on Half-Squat Training Volume and Repetition Performance in Strength-Trained Men: A Randomised Crossover Study
Brief Title: Post-activation Performance Enhancement Improves
Acronym: PAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Zarife Pancar, Associate Professor, University of Gaziantep
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GAUN-SBF-PANCAR-03; 2022/373 (Other: Clinical Research Local Ethics Committee)
Record Dates: First submitted 2025-02-04; First posted 2025-02-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-02

CONDITIONS: Resistance Exercise
Keywords: Post-Activation Performance; Resistance Training; Failure

STUDY DESIGN:
Intervention Model Description: This model is suitable because your study uses a randomized crossover design, where each participant undergoes both the PAPE and Control (CON) protocols in a randomized order, with a washout period between them to ensure full recovery.
Who Masked: Participant
Masking Description: This is a single-blind study where the participants are unaware of which protocol (PAPE or Control) they are assigned to during each session. The investigators who administer the protocols and measure the outcomes are also aware of the assignment. The randomization process is done prior to each session to determine the order of protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAPE Protocol (Experimental): Participants in this group will first perform a warm-up consisting of 3 repetitions at 90% of their 1RM. After a 10-minute rest, they will perform 3 sets of half-squats at 75% of their 1RM until volitional failure.
  Interventions: Behavioral: PAPE Protocol
- Control Protocol (Active Comparator): Participants in this group will perform a warm-up consisting of 8 repetitions at 50% of their 1RM. After a 4-minute rest, they will perform 3 sets of half-squats at 75% of their 1RM until volitional failure.
  Interventions: Behavioral: Control Protocol

INTERVENTIONS:
Behavioral: PAPE Protocol — In this intervention, participants perform a warm-up consisting of 3 repetitions at 90% of 1RM. After a 10-minute rest, they perform 3 sets of half-squats at 75% of their 1RM until volitional failure. This protocol is designed to enhance performance through the post-activation potentiation effect.
  Arms: PAPE Protocol
Behavioral: Control Protocol — In this intervention, participants perform a warm-up consisting of 8 repetitions at 50% of 1RM. After a 4-minute rest, they perform 3 sets of half-squats at 75% of their 1RM until volitional failure. This protocol is used as a baseline for comparison with the PAPE protocol.
  Arms: Control Protocol

SUMMARY:
This study investigates the acute effects of Post-Activation Performance Enhancement (PAPE) on the number of repetitions performed to volitional failure and total training volume in resistance-trained men. The research is designed as a randomized crossover trial where participants perform two different exercise protocols under controlled conditions.

The study includes 9 healthy, strength-trained male volunteers aged 18-30 years, with at least one year of resistance training experience. Participants complete two experimental conditions:

PAPE Protocol: A warm-up followed by 3 repetitions at 90% of 1RM, a 10-minute rest, and then 3 sets of half-squat at 75% 1RM until volitional failure.

Control (CON) Protocol: A warm-up followed by 8 repetitions at 50% of 1RM, a 4-minute rest, and then 3 sets of half-squat at 75% 1RM until volitional failure.

The primary outcome measures are:

Total training volume (set × reps × weight) Number of repetitions performed The study aims to determine whether PAPE improves total volume and repetition performance in resistance training. The findings could contribute to better training strategies for athletes and fitness professionals.

Ethical approval was obtained from the Gaziantep University Clinical Research Ethics Committee (Decision No: 2022/373), and all participants provided informed consent before participation.

DETAILED DESCRIPTION:
This study explores the acute effects of Post-Activation Performance Enhancement (PAPE) on repetition performance and training volume during a half-squat exercise in resistance-trained men. PAPE is a physiological phenomenon in which performance is enhanced following a conditioning activity (CA) involving a high-intensity resistance exercise. The study focuses on its effect on resistance training (RT) performance, specifically the number of repetitions performed to volitional failure and the total training volume during a half-squat exercise.

Study Design The study follows a randomized crossover design. Each participant performs both experimental protocols: PAPE and Control (CON) conditions. A random assignment is used to ensure that each participant experiences both conditions in separate sessions, with a 72-hour rest period between them to allow full recovery.

Participants Total number of participants: 9 trained male university students, aged 18-30 years, with at least 1 year of resistance training experience.

Inclusion Criteria:

Male participants aged 18-30 years No musculoskeletal disorders or injuries in the previous 6 months At least 1 year of continuous resistance training, including use of the half-squat exercise

Exclusion Criteria:

Doping or chronic drug use History of neuromuscular, metabolic, hormonal, or cardiovascular diseases Orthopedic limitations Use of supplements (e.g., caffeine) that may interfere with performance Participation in high-intensity training outside of the study protocol Interventions PAPE Protocol: Participants perform a warm-up consisting of 3 repetitions at 90% of 1RM, followed by a 10-minute rest. After the rest, they perform 3 sets of half-squats at 75% of 1RM until volitional failure.

Control (CON) Protocol: Participants perform a warm-up consisting of 8 repetitions at 50% of 1RM, followed by a 4-minute rest. After the rest, they perform 3 sets of half-squats at 75% of 1RM until volitional failure.

Outcome Measures

The primary outcomes of this study are:

Total Volume: The total weight lifted, calculated as set × repetitions × load. Repetition Count: The number of repetitions performed until volitional failure in each set.

Procedures Session 1: Anthropometric measurements are taken (e.g., height, weight, body mass index). Participants are familiarized with the half-squat exercise.

Session 2: 1RM (one-repetition maximum) for the half-squat is measured using a Smith machine.

Session 3 & 4: Participants are randomly assigned to either the PAPE or Control condition. Both protocols are performed on separate days, with 72 hours of rest in between.

Training and Testing Protocol Warm-Up: For PAPE, participants perform 3 repetitions at 90% of their 1RM. For the Control group, 8 repetitions at 50% of 1RM are performed.

Rest Periods: A 10-minute rest follows the PAPE warm-up, and a 4-minute rest follows the Control warm-up.

Testing Protocol: After the rest periods, participants perform 3 sets of half-squats at 75% of 1RM until failure in both conditions.

Ethical Considerations The study protocol has been approved by the Gaziantep University Clinical Research Ethics Committee (Decision No: 2022/373). All participants have provided written informed consent before their participation, ensuring their understanding of the study procedures and any potential risks.

Statistical Analysis Data will be analyzed using repeated measures ANOVA to compare total volume and repetition counts between the PAPE and Control conditions. Effect sizes will be calculated using Cohen's d for volume and partial eta-squared (ηp2) for repetition count.

Expected Impact This study aims to explore whether the PAPE protocol can significantly improve training outcomes by increasing the total volume and number of repetitions in a resistance training session, specifically in the half-squat exercise. If proven effective, PAPE could be incorporated into training strategies for athletes and fitness professionals aiming to maximize their performance and muscle hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18-30 years old.
* Only biologically male participants are eligible to participate in the study.
* Participants must have at least 1 year of continuous resistance training experience.
* Participants should be healthy, with no musculoskeletal disorders or injuries in the previous 6 months.
* Participants must have experience in performing the half-squat exercise as part of their regular training routine.
* Participants must be willing to provide written informed consent to participate in the study.

Exclusion Criteria:

* Participants who are currently using performance-enhancing drugs or have a history of chronic drug use.
* Participants with a history of neuromuscular disease, metabolic disorders, hormonal imbalances, cardiovascular diseases, or any orthopedic limitations.
* Participants who are using supplements such as caffeine or any other substances that might interfere with performance or the study protocol.
* Participants who perform high-intensity aerobic training or resistance training outside their routine, which may interfere with study procedures.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only individuals who self-identify as male are eligible to participate in this study. The study is limited to biological males, as all participants are required to be trained male athletes.
Enrollment: 9 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Total Training Volume (kg) | Immediately after exercise and 30 minutes post-exercise
  The total volume lifted during the half-squat exercise. It is calculated as set × repetitions × load for each set across all sets.

SECONDARY OUTCOMES:
Number of Repetitions Performed to Volitional Failure | Immediately after exercise and 30 minutes post-exercise
  The total number of repetitions performed to the point of volitional failure (when the participant can no longer perform the exercise).

CONTACTS AND LOCATIONS:
Overall Officials: Zarife Pancar Assistant Professor, PhD, Principal Investigator — University of Gaziantep
Locations (1):
- Gaziantep University, Faculty of Sport Sciences, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The following Individual Participant Data (IPD) will be shared after the completion of the study:
  Demographic Information: Age, sex, height, weight, and body mass index (BMI) for each participant.
  Training Data: Duration of resistance training experience and frequency of training per week.
  1RM Measurements: One-repetition maximum (1RM) values for the half-squat exercise for each participant.
  Outcome Measures:
  Total training volume (set × repetitions × load) during each protocol. Number of repetitions performed to volitional failure during each protocol. Fatigue Data: Self-reported fatigue levels after each set during the study. Protocol Data: Information on the exact sequence of protocols (PAPE vs. Control) that each participant underwent, including rest periods and exercise load.
  These data will be shared in anonymized form to ensure participant privacy and confidentiality. The data will be made available for future analysis or collaborations that support the study's aims, and will b
Supporting Information: Study Protocol, CSR
Time Frame: IPD and supporting information will be made available 6 months after the completion of data collection. The data will be accessible for 2 years following the publication of the study results, and will be shared with researchers upon request.
Access Criteria: Access will be provided electronically, through secure platforms like Data Access Repositories or institutional databases, with data being made available upon approval of the request.